CLINICAL TRIAL: NCT01187758
Title: Can Change in Physicians' Prescribing Habits Decrease Carriage of Resistant Bacteria in the Community?
Brief Title: Israeli Judicious Antibiotic Prescription Study
Acronym: IJAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Gili Regev-Yochay, Sheba medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-01-2357-GRY-CTIL
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Antibiotic Use; Carriage of Antibiotic Resistant Pathogens
Keywords: antibiotic use; antibiotic prescription; antibiotic resistant S. pneumoniae; MRSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational intervention (Experimental): Multifacet educational intervention that includes workshops, seminars and focus group meetings
  Interventions: Behavioral: Workshops and focus group meetings
- Control - no intervention (No Intervention): This group did not have any intervention, but their population was screened for carriage of antibiotic resistant bacteria

INTERVENTIONS:
Behavioral: Workshops and focus group meetings — Multifacet intervention that includes: Guideline preparation and implementation, preparing clinic campaign, improving knowledge about Ab resistance and diagnosis of respiratory infections
  Arms: Educational intervention

SUMMARY:
This study aims to implement judicious antibiotic prescription habits to primary care pediatricians using a multifacet educational intervention and assess two main outcomes: 1) Direct outcome - prescription rates of the physicians. 2)Indirect outcome - carriage of antibiotic resistant bacteria by the treated population, specifically nasopharyngeal S. pneumoniae, nasal S. aureus and rectal E.coli.

DETAILED DESCRIPTION:
Background: Bacterial antibiotic resistance is an increasing problem.

Aims: This study aims to implement judicious antibiotic prescription habits among 30 physicians and their treated population as compared to a control group of 30 physicians and their treated population. The outcomes to be measured are:

1. Change in antibiotic prescriptions to the treated patients of the intervention vs. control physicians during the study period (4years).
2. Change in carriage of antibiotic resistant pathogens, specifically nasopharyngeal penicillin resistant S. pneumoniae,nasal MRSA, and rectal quinolone resistant E. coli.

Study design: All primary care pediatricians of Hashfela district of Macabbi Healthcare services who will agree to participate will be randomly assigned to an intervention or control group. The intervention group will be led by local leaders (primary care physicians from that district) and will take part in educational activities involving annual workshops and quarterly focus group meetings. The intervention is a multifacet intervention that will include guideline preparation, knowledge building, dealing with uncertainties, etc.

The patients of both intervention and control physicians will be screened twice a year for carriage of the bacteria mentioned above. Cross-sectional screening of the treated population will be carried in Summer and winter for 5 consecutive years. Screening will include signing an informed consent, filling a questionnaire and screening with nasal, nasopharyngeal and rectal swabs.

ELIGIBILITY:
Inclusion Criteria:

* All treated patients of the participating physicians under the age of 5y, who came for any reason for a visit during the study period, who's parents agreed to participate.

Exclusion Criteria:

The only reason to exclude a child from being recruited was age>5y or refusal of the parent/child to participate.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5700 (Actual)
Dates: Start 2002-02; Primary Completion 2005-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
antibiotic prescription rate of physicians | 5 years
  Antibiotic prescrption rate at baseline will be compared to changes following the intervention between the 2 groups (control and intervention).

SECONDARY OUTCOMES:
Carriage of antibiotic resistant bacteria by treated patients | 4 years
  Every summer and winter a crosssectional survey of the treated patients of the control and intervention physicians will be carried out to determine the rate of carriage of penicillin-resistant S. pneumonaie, MRSA and Quinolone-resistant E.coli.

REFERENCES:
- [Derived] Regev-Yochay G, Raz M, Dagan R, Roizin H, Morag B, Hetman S, Ringel S, Ben-Israel N, Varon M, Somekh E, Rubinstein E. Reduction in antibiotic use following a cluster randomized controlled multifaceted intervention: the Israeli judicious antibiotic prescription study. Clin Infect Dis. 2011 Jul 1;53(1):33-41. doi: 10.1093/cid/cir272. PMID 21653300